CLINICAL TRIAL: NCT05037487
Title: Evaluation of Smoked THC and CBD in Oral Fluid, Pharmacokinetics, and Subjective and Neurocognitive Effects in Men and Women
Brief Title: Evaluation of Smoked THC and CBD in Men and Women
Acronym: S-TACOFS
Status: Recruiting | Phase: Phase 1 | Type: Interventional
Sponsor: University of California, Los Angeles (Other)
Responsible Party: Principal Investigator, Ziva D. Cooper, PhD, Associate Professor, University of California, Los Angeles
Allocation: Randomized | Model: Crossover | Masking: Double | Purpose: Basic Science
Other Study IDs: 21-001137
Record Dates: First submitted 2021-08-31; First posted 2021-09-08 (Actual); Last update posted 2025-04-04 (Actual); Status verified 2024-07

CONDITIONS: Drug Abuse; Intoxication by Drug; Impairment
Keywords: Cannabis; THC; CBD; Intoxication; Impairment
MeSH Terms: conditions — Substance-Related Disorders; Marijuana Abuse

STUDY DESIGN:
Intervention Model Description: This is a randomized, double-blind, placebo-controlled study. All participants will complete all dose conditions in a randomized order.
Who Masked: Participant, Investigator
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: Yes | FDA-regulated Device: No | US Export: No

ARMS (4):
- Placebo (Placebo Comparator): Smoked placebo cannabis
  Interventions: Drug: Placebo Cannabis
- 20 mg CBD (Experimental): Smoked cannabis with CBD
  Interventions: Drug: 20 mg CBD Cannabis
- 20 mg CBD + 20 mg THC (Experimental): Smoked cannabis with CBD and THC
  Interventions: Drug: 20 mg CBD + 20 mg THC Cannabis
- 20 mg THC (Experimental): Smoked cannabis with THC
  Interventions: Drug: 20 mg THC Cannabis

INTERVENTIONS:
Drug: Placebo Cannabis — Smoked placebo cannabis
  Arms: Placebo
Drug: 20 mg CBD Cannabis — Smoked cannabis with CBD
  Arms: 20 mg CBD
Drug: 20 mg CBD + 20 mg THC Cannabis — Smoked cannabis with CBD and THC
  Arms: 20 mg CBD + 20 mg THC
Drug: 20 mg THC Cannabis — Smoked cannabis with THC
  Arms: 20 mg THC

SUMMARY:
The purpose of this study is to determine the pharmacokinetics and pharmacodynamics of inhaled cannabis with varying amounts of delta-9-tetrahydrocannabinol (THC), and cannabidiol (CBD) and to evaluate detection of recently smoked THC in oral fluid.

DETAILED DESCRIPTION:
This double-blind placebo controlled, within-subject study study will assess testing devices that can measure biochemical markers in oral fluid and neurocognitive-performance markers of recent cannabis use. Other pharmacodynamic effects of inhaled cannabis with CBD and THC will be determined and the pharmacokinetics of THC, CBD, and respective metabolites will be assessed in whole blood.

ELIGIBILITY:
Inclusion Criteria:

* Male or non-pregnant and non-lactating females aged 21-55 years
* Report weekly-monthly use of cannabis (≤1 day per week) over the past month prior to screening,
* Not currently seeking treatment for their cannabis use
* Have a Body Mass Index from 18.5 - 34kg/m2.
* Able to perform all study procedures
* Must be using a contraceptive (hormonal or barrier methods)

Exclusion Criteria:

* Meeting DSM-V criteria for moderate to severe Cannabis Use disorder (CUD) or any substance use disorder other than nicotine, caffeine
* Any other Axis I disorder
* Report using other illicit drugs in the prior 4 weeks, other than cannabis.
* Current use of any medications that may affect study outcomes
* If medical history, physical and psychiatric examination, or laboratory tests performed during the screening process are not within the normal range and / or reveal any significant illness (e.g., hypertension) as judged by the study physician and to put the participant at greater risk of experiencing adverse events due to completion of study procedures.
* Pregnancy is exclusionary due to the possible effects of the study medication on fetal development.
* History of an allergic reaction or adverse reaction to cannabis is exclusionary.
* History of respiratory illness or current respiratory illness
* Currently enrolled in another research protocol
* Not using a contraceptive method (hormonal or barrier methods)
* The evaluating physician reviews all medical assessments along with medical history. Any disorders that might make cannabis administration hazardous are exclusionary.

Ages: 21 Years to 55 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Adult
Enrollment: 22 (Estimated)
Dates: Start 2022-09-01 (Actual); Primary Completion 2025-09-01 (Estimated); Study Completion 2026-09-01 (Estimated)

PRIMARY OUTCOMES:
Subjective drug effect ratings of impairment and abuse liability | 6 hours
  Peak subjective ratings of drug effects associated with abuse liability and impairment as measured using visual analogue scales (VAS; 1-100mm).
Pharmacokinetics of THC, CBD and metabolites | 6 hours
  Peak blood levels of THC, CBD, 11-OH-THC, and THCCOOH after exposure (Tmax)
Behavioral task performance as assessed by the DRUID App Score | 6 hour
  Trough composite scores on the DRUID App
THC concentrations in oral fluid | 6 hour
  Peak levels of THC in oral fluid after exposure

CONTACTS AND LOCATIONS:
Overall Officials: Ziva Cooper, PhD, Principal Investigator — University of California, Los Angeles
Locations (1):
- University of California, Los Angeles, Los Angeles, California, United States

IPD SHARING:
Plan to Share IPD: No